CLINICAL TRIAL: NCT02611804
Title: A Randomized, Double-Blind, Parallel-Group, Vehicle-Controlled, Multicenter Study Comparing Diclofenac Sodium Gel, 3% to Solaraze® Gel, 3% in the Treatment of Actinic Keratosis on the Face or Bald Scalp
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: SYM 2015-01
Record Dates: First submitted 2015-11-19; First posted 2015-11-23 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic | interventions — Diclofenac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Diclofenac Sodium Gel, 3% (Experimental): Diclofenac Sodium Gel, 3%, applied twice daily for 60 days
  Interventions: Drug: Diclofenac sodium
- Solaraze® (Active Comparator): Solaraze® (diclofenac sodium) Gel, 3%, applied twice daily for 60 days
  Interventions: Drug: Diclofenac sodium
- Vehicle of Test Product (Placebo Comparator): Vehicle of Test Product, Gel, applied twice daily for 60 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Diclofenac sodium
  Arms: Diclofenac Sodium Gel, 3%
Drug: Diclofenac sodium
  Other Names: Solaraze®
  Arms: Solaraze®
Drug: Placebo
  Arms: Vehicle of Test Product

SUMMARY:
To compare the efficacy and safety profiles of Teva's Diclofenac Sodium Gel, 5% (test product) to Solaraze® (diclofenac sodium) Gel, 3% (reference product) to demonstrate the clinical equivalence and to show that the efficacy of the 2 active formulations is superior to that of vehicle in treating subjects with actinic keratosis (AK) on the face or bald scalp.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent for the study.
* At least 18 years of age
* Immunocompetent male or nonpregnant and nonlactating female. Each female subject of childbearing potential (excluding women who are surgically sterilized or postmenopausal for at least 2 years), in addition to having a negative urine pregnancy test at Visit 1/Day 1, must be willing to use an acceptable form of birth control during the study. For the purpose of this study, the following are considered acceptable methods of birth control: oral contraceptives, contraceptive patches, contraceptive implant, vaginal contraceptive, double-barrier methods (e.g., condom and spermicide), contraceptive injection (Depo-Provera®), intrauterine device IUD (Mirena®), Essure®, and abstinence with a documented second acceptable method of birth control if the subject becomes sexually active.
* Clinical diagnosis of AK, defined as ≥ 5 and ≤ 10 clinically typical, visible, discrete, nonhyperkeratotic, nonhypertrophic AK lesions, each at least 4 mm in diameter, contained within a 25-cm2 treatment area on either the face or bald scalp, but not both face and scalp.
* In general good health and free from any clinically significant disease, other than AK, that might interfere with the study evaluations.
* Willing and able to understand and comply with the requirements of the study, apply the study medication as instructed, attend the required visits, comply with therapy prohibitions, and be able to complete the study.

Exclusion Criteria:

* Presence of active gastrointestinal ulceration or bleeding.
* Presence of severe renal or hepatic impairment.
* Presence of atopic dermatitis, basal cell carcinoma, eczema, psoriasis, rosacea, squamous cell carcinoma, sunburn, or other possible confounding skin conditions on the treatment area of either the face or bald scalp.
* Clinically significant systemic disease (immunological deficiencies), unstable medical disorder, life-threatening disease, or current malignancies.
* Use within 6 months (180 days) prior to randomization of oral isotretinoin.
* Use within 6 months (180 days) prior to randomization on the face or bald scalp where the designated treatment area is located of 1) chemical peel, 2) dermabrasion, 3) laser abrasion, 4) PUVA (psoralen plus ultraviolet A) therapy, or 5) UVB therapy.
* Use within 6 months (180 days) prior to randomization of systemic cancer chemotherapy medications.
* Use within 1 month (30 days) prior to randomization on the face of bald scalp where the designated treatment are is located of 1) cryodestruction or chemodestruction, 2) curettage, 3) photodynamic therapy, 4) surgical excision, 5) topical 5-fluorouracil, 6) topical corticosteroids, 7) topical diclofenac, 8) topical imiquimod, 9) topical retinoids, 10) other treatments for actinic keratosis.
* Use within 1 month (30 days) prior to randomization of 1) immunomodulators or immunosuppressive therapies, 2) interferon, 3) systemic (oral and injectable) corticosteroids, 4) cytotoxic drugs. Intranasal or inhaled corticosteroids are acceptable if kept constant throughout the study. Intra-articular injection of steroids is acceptable for this study.
* Known hypersensitivity or allergies to diclofenac, benzyl alcohol, polyethylene glycol monomethyl ether 359, hyaluronate sodium or any component of the study medication (in any dosage form).
* Previous or current history of allergies to aspirin (ASA) or other NSAIDS.
* Females who are pregnant, breastfeeding, intending to become pregnant during the study, or who do not agree to use an acceptable form of birth control during the study.
* Any clinically significant condition or situation other than the condition being studied that, in the opinion of the investigator, would interfere with the study evaluation or optimal participation in the study.
* Use of any investigational drug or investigational device within 1 month (30 days) prior to the randomization.
* Previous participation in this study.
* Current involvement in activities that require excessive or prolonged sun exposure.
* Consumption of excessive alcohol, abuse of drugs, or a condition that could compromise the subject's ability to comply with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 492 (Actual)
Dates: Start 2015-10; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Proportion of Patients with Treatment Success at Visit 4 | Day 90

CONTACTS AND LOCATIONS:
Locations (30):
- United States (30):
  - Agave Clinical Research, Mesa, Arizona
  - Radiant Research, Inc., Tucson, Arizona
  - Center for Dermatology Clinical Research, Inc., Fremont, California
  - Medical Center for Clinical Research, San Diego, California
  - TCR Medical Corporation, San Diego, California
  - Clinical Science Institute, Santa Monica, California
  - Horizons Clinical Research Center, Denver, Colorado
  - Olympian Clinical Research, Clearwater, Florida
  - Tampa Bay Medical Research, Clearwater, Florida
  - Renstar Medical Research, Ocala, Florida
  - DS Research, Louisville, Kentucky
  - Dermatology Consulting Services, High Point, North Carolina
  - DermOne of North Carolina, Wilmington, North Carolina
  - PMG Research of Winston-Salem, Winston-Salem, North Carolina
  - Radiant Research, Cincinnati, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Omega Medical Research, Warwick, Rhode Island
  - Radiant Research, Anderson, South Carolina
  - Greenville Dermatology, Greenville, South Carolina
  - Dermatology Associates of Knoxville, Knoxville, Tennessee
  - The Skin Wellness Center, Knoxville, Tennessee
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - DermResearch, Inc., Austin, Texas
  - The Center for Skin Research, Houston, Texas
  - ACRC Trials, Plano, Texas
  - Dermatology Clinical Research Center of San Antonio, San Antonio, Texas
  - Stephen Miller, M.D., San Antonio, Texas
  - Dermatology Research Center, Salt Lake City, Utah
  - The Education and Research Foundation, Lynchburg, Virginia
  - Premier Clinical Research, Spokane, Washington